CLINICAL TRIAL: NCT02685540
Title: Death Rate in Anesthesia: A Retrospective Study of Five Years Period From a Tertiary Hospital
Brief Title: Death Rate in Anesthesia: A Study in a Tertiary Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Subhi M. Alghanem, Professor of Anesthesia and Intensive Care, University of Jordan
Other Study IDs: 190/14a/tk
Record Dates: First submitted 2016-02-14; First posted 2016-02-18 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Sudden Death
Keywords: Anesthesia; mortality
MeSH Terms: conditions — Death, Sudden

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Death rate in anesthesia is one of the most valuable methods to assess the safety of anesthesia practice among different types of patients.

In the investigators study, the investigator will review the death rate in anesthesia whether regional or general over the past five years from 2010 to 2014, by examining the patients records from the hospital database.

DETAILED DESCRIPTION:
Death rate in anesthesia is one of the most valuable methods to assess the safety of anesthesia practice among different types of patients. Most of the studies of death rate in anesthesia are retrospective. Although retrospective studies suffer many draw backs in their design and results, but they are still common method to evaluate the safety of anesthesia practice for surgical patients.

In the investigators study, the investigators will review the death rate in anesthesia whether regional or general over the past five years from 2010 to 2014, by examining the patients records from the hospital database.

The cause of death will be grouped into: totally anesthesia related, partially anesthesia related, surgery related or patient condition related.

The records and files of dead patients will be examined by committee from the researchers to estimate the cause of death.

The end point of the investigators study will be anesthesia death rate inside the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent anesthesia and surgery.
* Patients who died inside the hospital.

Exclusion Criteria:

* Patient who underwent anesthesia and surgery and do not died and discharged home.
* Patients who died outside the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent anesthesia and surgery and died inside the hospital
Sampling Method: Non-Probability Sample
Enrollment: 792 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
number of anesthetized patients who died in the perioperative period inside the hospital | 30 days post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Subhi M Alghanem, FFARCS, Study Chair — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watters DA, Hollands MJ, Gruen RL, Maoate K, Perndt H, McDougall RJ, Morriss WW, Tangi V, Casey KM, McQueen KA. Perioperative mortality rate (POMR): a global indicator of access to safe surgery and anaesthesia. World J Surg. 2015 Apr;39(4):856-64. doi: 10.1007/s00268-014-2638-4. PMID 24841805